CLINICAL TRIAL: NCT05527340
Title: Multicenter, Phase II, National and Open-label Study to Evaluate Iberdomide-dexamethasone Alone or in Combination With Standard MM Treatment Regimens in Transplant Ineligible Newly Diagnosed Patients.
Brief Title: Iberdomide-dexamethasone Alone or in Combination With Standard MM Treatment Regimens in Transplant Ineligible Newly Diagnosed Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Celgene-BMS (Unknown); Janssen-Cilag, S.A. (Industry); LIDESEC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-IBERDARAX; 2021-002190-25 (EudraCT Number)
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: De novo Multiple Myeloma; Transplant ineligible
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iberdomide + dexamethasone (IBERDEX) (Experimental): IBERDEX
  * Iberdomide on days 1 to 21 at 1.6 mg, every 4 weeks, orally (PO).
  * Dexamethasone will be given on days 1, 8, 15, and 22 at 40 mg (patients aged ≥ 75 years: 20 mg), every 4 weeks, PO.
  Interventions: Drug: Iberdomide; Drug: Dexamethasone
- iberdomide + daratumumab + dexamethasone (IBERDARADEX) (Experimental): IBERDARADEX
  * Iberdomide on days 1 to 21 at 1.6 mg, every 4 weeks, PO.
  * Dexamethasone will be given on days 1, 8, 15, and 22 at 40 mg (patients aged ≥ 75 years: 20 mg), every 4 weeks, PO.
  * Daratumumab will be given at 1800 mg, every 4 weeks, subcutaneously (SC). Cycles 1 and 2 (C1 and C2): Days 1, 8, 15, and 22 C3-6: Days 1 and 15 From C7 onwards: Day 1 of each cycle Cycles will be of 4 weeks of duration (28 days).
  Interventions: Drug: Iberdomide; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Iberdomide — Iberdomide on days 1 to 21 at 1.6 mg, every 4 weeks, orally (PO)
Drug: Dexamethasone — Dexamethasone 40 mg (PO) (or 20 mg (PO) if patient ≥ 75 years old) should be administered on the days 1, 8, 15 and 22 of every 4-week cycle.
Drug: Daratumumab — Daratumumab will be given at 1800 mg, every 4 weeks, subcutaneously (SC). Cycles 1 and 2 (C1 and C2): Days 1, 8, 15, and 22 C3-6: Days 1 and 15 From C7 onwards: Day 1 of each cycle Cycles will be of 4 weeks of duration (28 days).
  Arms: iberdomide + daratumumab + dexamethasone (IBERDARADEX)

SUMMARY:
This is a multicenter, phase II, national, and open-label study to evaluate the efficacy and safety of two different combinations, iberdomide-dexamethasone (IBERDEX) and iberdomide-dexamethasone in combination with daratumumab (IBERDARADEX) in transplant ineligible newly diagnosed multiple myeloma (NDMM) patients. It will be ensured that at least 30% of the patients are frail in order to evaluate the feasibility of these combinations in this special population.

Patients will receive treatment with either iberdomide + dexamethasone (IBERDEX) or iberdomide + daratumumab + dexamethasone (IBERDARADEX), until unacceptable toxicity, disease progression, patient withdrawal, loss to follow-up, end of study or death, whichever comes first. This is not a randomized trial so eligible patients will be sequentially allocated to receive iberdomide-dexamethasone or iberdomide-dexamethasone plus daratumumab.

DETAILED DESCRIPTION:
This is a multicenter, phase II, national, and open-label study to evaluate the efficacy and safety of two different combinations, iberdomide-dexamethasone (IBERDEX) and iberdomide-dexamethasone in combination with daratumumab (IBERDARADEX) in transplant ineligible newly diagnosed multiple myeloma (NDMM) patients. It will be ensured that at least 30% of the patients are frail in order to evaluate the feasibility of these combinations in this special population.

Patients will receive treatment with either iberdomide + dexamethasone (IBERDEX) or iberdomide + daratumumab + dexamethasone (IBERDARADEX), until unacceptable toxicity, disease progression, patient withdrawal, loss to follow-up, end of study or death, whichever comes first. This is not a randomized trial so eligible patients will be sequentially allocated to receive iberdomide-dexamethasone or iberdomide-dexamethasone plus daratumumab.

Participants will be evaluated for study eligibility per protocol as defined in the Inclusion/Exclusion criteria . The screening period takes place 28 days prior to the baseline visit.

Frontline treatment: cohorts 1 and 2

Cohort 1: IBERDEX

* Iberdomide on days 1 to 21 at 1.6 mg, every 4 weeks, orally (PO).
* Dexamethasone will be given on days 1, 8, 15, and 22 at 40 mg (patients aged ≥ 75 years: 20 mg), every 4 weeks, PO.

Cohort 2: IBERDARADEX

* Iberdomide on days 1 to 21 at 1.6 mg, every 4 weeks, PO.
* Dexamethasone will be given on days 1, 8, 15, and 22 at 40 mg (patients aged ≥ 75 years: 20 mg), every 4 weeks, PO.
* Daratumumab will be given at 1800 mg, every 4 weeks, subcutaneously (SC). Cycles 1 and 2 (C1 and C2): Days 1, 8, 15, and 22 C3-6: Days 1 and 15 From C7 onwards: Day 1 of each cycle

The study treatment in both cohorts will be until unacceptable toxicity, disease progression, patient withdrawal, loss to follow-up, end of study or death, whichever comes first.

The trial has the following objectives:

Primary Objectives

PO1: To determine the efficacy of iberdomide in combination with dexamethasone (IBERDEX cohort 1) and also in combination with daratumumab and dexamethasone (IBERDARADEX cohort 2) in transplant ineligible NDMM patients, as measured by overall response rate (ORR) as well as the other response categories and especially the complete response rate (CRR) according to the International Myeloma Working Group (IMWG) response criteria 2016.

Secondary Objectives

SO1: To evaluate the efficacy in terms of minimal residual disease (MRD) with especial attention to the proportion of patients in MRD negative at 12 months of starting treatment as well as patients able to sustain it over time (according to the IMWG response criteria 2016).

SO2: To evaluate time to event data in the overall population and in the frail and non-frail population: Progression Free Survival (PFS) (from the time of inclusion in the trial until progression and/or death) and Overall Survival (OS).

SO3: To evaluate the changes in the immune profiling in order to better understand the outcomes in the overall population and in the non-frail and frail subgroups of patients.

SO4: To assess quality of life evolution through EQ-5D/5L, QLQ-C30 and MY20 questionnaires, at baseline and at months 4, 8, 12, 18, and 24.

SO5: To assess the safety of the combination of iberdomide + dexamethasone and iberdomide + dexamethasone + daratumumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
2. Patient must be able to understand the study procedures.
3. Patient has given voluntary written informed consent before performance of any study-related procedure nor part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
4. Newly diagnosed multiple myeloma patient ≥65 years or younger but non-transplant eligible who requires start active treatment according to the IMWG published in 2014.
5. Patient must have a measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200 mg/24 h. For patients whose disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/L (100 mg/dl), with an abnormal serum FLC ratio.
6. Patient is defined as non-frail or frail using the modified-IMWG scale (APPENDIX 5). Frailty score according to the modified-IMWG scale will be collected before starting the treatment in order to ensure 30% of the patients are frail.
7. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
8. Patient must be ≥ 18 years of age
9. Patient must have adequate organ function,
10. Female childbearing potential patient (FCBP) criteria: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    A female patient is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
    * Is not a female of childbearing potential (FNCBP) OR
    * Is a FCBP and

      * She understands the potential teratogenic risk to the unborn child
      * She understands the need for effective contraception, without interruption, 28 days before starting study treatment, throughout the entire duration of study treatment, during dose interruptions and for at least 3 months after the last dose of study treatment.
      * She understands and agrees to inform the Investigator if a change or stop of method of contraception is needed
      * She must be capable of complying with effective contraceptive measures
      * She is informed and understands the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
      * She understands the need to commence study treatment as soon as it is dispensed following a negative pregnancy test
      * She understands and accepts the need to undergo pregnancy testing based on the frequency outlined in this plan
      * She acknowledges she understands the hazards study drugs can cause to an unborn fetus and the necessary precautions associated with the use of study drugs.

    The Investigator must ensure that a FCBP:
    * Complies with the conditions of the pregnancy prevention plan, including confirmation that she has an adequate level of understanding
    * Acknowledges the aforementioned requirements. A FCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 24 hours before the first dose of study drug(s).

    Non-childbearing potential is defined as follows (by other than medical reasons):
    * Has not achieved menarche at some point
    * Has undergone a hysterectomy or bilateral oophorectomy
    * Has been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
11. Male patient: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    Male patient is eligible to participate if he agrees to the following during dose interruptions and for at least 3 months following the last dose of iberdomide to allow for clearance of any altered sperm:
    * Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a FCBP
    * Understand the need for the use of a condom even if he has had a vasectomy, if engaged in sexual activity with a pregnant female or a FCBP
    * Understand the potential teratogenic risk if the subject donates semen or sperm.
    * Understand that the effects on fertility are currently unknown, therefore all family planning options and/or alternatives should be thoroughly discussed with the study doctor prior to receiving study drugs.
12. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0 must be ≤ Grade 1 at the time of enrolment except for alopecia

Exclusion Criteria:

1. Patient has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia or active POEMS syndrome at the time of screening.
2. Patient has had clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS multiple myeloma.
3. Patient has invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
4. Any serious medical condition that places the subject at an unacceptable risk if he or she participates in this study; subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
5. Pregnant or breastfeeding females.
6. Patient is simultaneously enrolled in other interventional clinical trial.
7. Received plasmapheresis within 7 days prior to the first dose of study drug.
8. Patient has received prior radiotherapy within 2 weeks of start of study therapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
9. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to iberdomide or drugs chemically related to iberdomide, or any of the excipients contained in the formulation of the study treatment.
10. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to daratumumab or drugs chemically related to daratumumab, or any of the excipients contained in the formulation of the study treatment.
11. Participant has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to other monoclonal antibodies.
12. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to dexamethasone or drugs chemically related to dexamethasone, or any of the excipients contained in the formulation of the study treatment.
13. Major surgery (except kyphoplasty) ≤ 4 weeks prior to initiating protocol therapy.
14. Patient has peripheral neuropathy or neuropathic pain grade ≥2, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTC AE) Version 5.0.
15. Patient evidence of cardiovascular risk including any of the following:

    * QTcF interval QTcF > 480 msec (the QT interval values must be corrected for heart rate by Fridericia's formula [QTcF])
    * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening.
    * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
    * Uncontrolled hypertension, defined as an average systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg despite optimal treatment.
16. Patient has current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
17. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect patient's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria
18. Evidence of active mucosal or internal bleeding.
19. Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.
20. Uncontrolled endocrine diseases (i.e. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
21. Patients with acute diffuse infiltrative pulmonary disease and/or pericardial disease.
22. Patients with severe chronic obstructive pulmonary disease (COPD) or asthma with forced expiratory volume in the first minute (FEV1) less than 50%.
23. History of interstitial lung disease or ongoing interstitial lung disease.
24. Patient has an active infection requiring antibiotic, antiviral, or antifungal treatment
25. Participant has known HIV infection
26. Patient has presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment.

aa.Patient has positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.

Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Throught the study period. Approximately 6 years.
  The percentage of participants with a confirmed partial response (PR) or better (PR, Very good partial response (VGPR), Complete response (CR), stringent complete response (sCR)).Response rates will be monitored monthly, but the study will report the % of patients achieving CR rate at month 12, 18, 24 and yearly thereafter.
Complete Response Rate (CRR) | Throught the study period. Approximately 6 years.
  The percentage of participants with a confirmed complete response (CR) or better (stringent complete response (CR, sCR).

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negativity rate | Throught the study period. Approximately 6 years.
  The percentage of participants who are MRD negative by next-generation flow cytometry (NGF), PET/CT, and mass spectrometry.
Progression-Free Survival (PFS) | Throught the study period. Approximately 6 years.
  Time from the date of randomization until the earliest date of documented disease progression or death due to any cause.
Overall Survival (OS) | Throught the study period. Approximately 6 years.
  Time from the date of randomization until the date of death due to any cause
Changes in the immune profiling. | Throught the study period. Approximately 6 years.
  Relative distribution and immunophenotype of inmune profiling from baseline onto treatment, remission and disease progression.
Health status/quality of life | Baseline and throught the first 24 months.
  Global health status/quality of life based on patient reported outcome: EQ-5D/5L questionnaire.
Health status/quality of life | Baseline and throught the first 24 months.
  Global health status/quality of life based on patient reported outcome: QLQ-C30 questionnaire.
Health status/quality of life | Baseline and throught the first 24 months.
  Global health status/quality of life based on patient reported outcome: MY20 questionnaire.
Frequency and percentage of deaths and primary cause of death. | Throught the study period. Approximately 6 years.
  Incidence of deaths and primary cause of death for safety analysis.
Incidence of adverse events (AEs). | Throught the treatment period. Approximately 4 years.
  Incidence of adverse events (AEs).
Percentage of patients discontinuing therapy due to AEs. | Throught the treatment period. Approximately 4 years.
  Percentage of patients discontinuing therapy due to AEs.
Percentage of patients requiring dose modifications. | Throught the treatment period. Approximately 4 years.
  Percentage of patients requiring dose modifications.
Percentage of patients with changes in laboratory analytes from the hematology and blood chemistry panel. | Throught the treatment period. Approximately 4 years.
  Percentage of patients with changes in laboratory analytes from the hematology and blood chemistry panel.

CONTACTS AND LOCATIONS:
Overall Officials: María Victoria Mateos Manteca, Study Chair — University of Salamanca; Verónica González de la Calle, Study Chair — University of Salamanca; Jesús San Miguel Izquierdo, Study Chair — Clínica Universidad de Navarra; Juan José Lahuerta Palacios, Study Chair — Hospital Universitario 12 de Octubre; Joan Bladé Creixenti, Study Chair — Hospital Clinic of Barcelona
Locations (9):
- Spain (9):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe de Valencia, Valencia

REFERENCES:
- [Background] Mateos MV, San Miguel JF. Management of multiple myeloma in the newly diagnosed patient. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):498-507. doi: 10.1182/asheducation-2017.1.498. PMID 29222298
- [Background] Durie BGM, Kumar SK, Usmani SZ, Nonyane BAS, Ammann EM, Lam A, Kobos R, Maiese EM, Facon T. Daratumumab-lenalidomide-dexamethasone vs standard-of-care regimens: Efficacy in transplant-ineligible untreated myeloma. Am J Hematol. 2020 Dec;95(12):1486-1494. doi: 10.1002/ajh.25963. Epub 2020 Sep 5. PMID 32804408
- [Background] Belotti A, Ribolla R, Cancelli V, Crippa C, Bianchetti N, Ferrari S, Bottelli C, Cattaneo C, Tucci A, De La Fuente Barrigon C, Rossi G. Transplant eligibility in elderly multiple myeloma patients: Prospective external validation of the international myeloma working group frailty score and comparison with clinical judgment and other comorbidity scores in unselected patients aged 65-75 years. Am J Hematol. 2020 Jul;95(7):759-765. doi: 10.1002/ajh.25797. Epub 2020 Apr 23. PMID 32242970
- [Background] Facon T, Dimopoulos MA, Meuleman N, Belch A, Mohty M, Chen WM, Kim K, Zamagni E, Rodriguez-Otero P, Renwick W, Rose C, Tempescul A, Boyle E, Manier S, Attal M, Moreau P, Macro M, Leleu X, Lorraine Chretien M, Ludwig H, Guo S, Sturniolo M, Tinel A, Silvia Monzini M, Costa B, Houck V, Hulin C, Yves Mary J. A simplified frailty scale predicts outcomes in transplant-ineligible patients with newly diagnosed multiple myeloma treated in the FIRST (MM-020) trial. Leukemia. 2020 Jan;34(1):224-233. doi: 10.1038/s41375-019-0539-0. Epub 2019 Aug 19. PMID 31427722
- [Background] Cruz-Jentoft AJ, Gonzalez B, de la Rubia J, Hernandez Rivas JA, Soler JA, Fernandez Lago C, Arnao M, Gironella M, Perez Persona E, Zudaire MT, Olivier C, Altes A, Garcia Guinon A, Nomdedeu B, Arnan M, Ramirez Payer A, Sanchez-Godoy P, Pajuelo N, Vilanova D, Monjil DF, Bonanad S; GAH Group. Further psychometric validation of the GAH scale: Responsiveness and effect size. J Geriatr Oncol. 2017 May;8(3):211-215. doi: 10.1016/j.jgo.2016.12.008. Epub 2016 Dec 22. PMID 28017687
- [Background] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Komarnicki M, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Lisby S, Khokhar NZ, O'Rourke L, Chiu C, Qin X, Guckert M, Ahmadi T, Moreau P; POLLUX Investigators. Daratumumab, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Oct 6;375(14):1319-1331. doi: 10.1056/NEJMoa1607751. PMID 27705267
- [Background] Bahlis NJ, Dimopoulos MA, White DJ, Benboubker L, Cook G, Leiba M, Ho PJ, Kim K, Takezako N, Moreau P, Kaufman JL, Krevvata M, Chiu C, Qin X, Okonkwo L, Trivedi S, Ukropec J, Qi M, San-Miguel J. Daratumumab plus lenalidomide and dexamethasone in relapsed/refractory multiple myeloma: extended follow-up of POLLUX, a randomized, open-label, phase 3 study. Leukemia. 2020 Jul;34(7):1875-1884. doi: 10.1038/s41375-020-0711-6. Epub 2020 Jan 30. PMID 32001798
- [Background] Dimopoulos MA, San-Miguel J, Belch A, White D, Benboubker L, Cook G, Leiba M, Morton J, Ho PJ, Kim K, Takezako N, Moreau P, Kaufman JL, Sutherland HJ, Lalancette M, Magen H, Iida S, Kim JS, Prince HM, Cochrane T, Oriol A, Bahlis NJ, Chari A, O'Rourke L, Wu K, Schecter JM, Casneuf T, Chiu C, Soong D, Sasser AK, Khokhar NZ, Avet-Loiseau H, Usmani SZ. Daratumumab plus lenalidomide and dexamethasone versus lenalidomide and dexamethasone in relapsed or refractory multiple myeloma: updated analysis of POLLUX. Haematologica. 2018 Dec;103(12):2088-2096. doi: 10.3324/haematol.2018.194282. Epub 2018 Sep 20. PMID 30237262
- [Background] Facon T, Kumar S, Plesner T, Orlowski RZ, Moreau P, Bahlis N, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, O'Dwyer M, Perrot A, Venner CP, Weisel K, Mace JR, Raje N, Attal M, Tiab M, Macro M, Frenzel L, Leleu X, Ahmadi T, Chiu C, Wang J, Van Rampelbergh R, Uhlar CM, Kobos R, Qi M, Usmani SZ; MAIA Trial Investigators. Daratumumab plus Lenalidomide and Dexamethasone for Untreated Myeloma. N Engl J Med. 2019 May 30;380(22):2104-2115. doi: 10.1056/NEJMoa1817249. PMID 31141632
- [Background] Perrot A, Facon T, Plesner T, Usmani SZ, Kumar S, Bahlis NJ, Hulin C, Orlowski RZ, Nahi H, Mollee P, Ramasamy K, Roussel M, Jaccard A, Delforge M, Karlin L, Arnulf B, Chari A, He J, Ho KF, Van Rampelbergh R, Uhlar CM, Wang J, Kobos R, Gries KS, Fastenau J, Weisel K. Health-Related Quality of Life in Transplant-Ineligible Patients With Newly Diagnosed Multiple Myeloma: Findings From the Phase III MAIA Trial. J Clin Oncol. 2021 Jan 20;39(3):227-237. doi: 10.1200/JCO.20.01370. Epub 2020 Dec 16. PMID 33326255
- [Background] Ito T, Handa H. [Cereblon as a primary target of IMiDs]. Rinsho Ketsueki. 2019;60(9):1013-1019. doi: 10.11406/rinketsu.60.1013. Japanese. PMID 31597822
- [Background] Bjorklund CC, Kang J, Amatangelo M, Polonskaia A, Katz M, Chiu H, Couto S, Wang M, Ren Y, Ortiz M, Towfic F, Flynt JE, Pierceall W, Thakurta A. Iberdomide (CC-220) is a potent cereblon E3 ligase modulator with antitumor and immunostimulatory activities in lenalidomide- and pomalidomide-resistant multiple myeloma cells with dysregulated CRBN. Leukemia. 2020 Apr;34(4):1197-1201. doi: 10.1038/s41375-019-0620-8. Epub 2019 Nov 12. No abstract available. PMID 31719682
- [Background] Matyskiela ME, Zhang W, Man HW, Muller G, Khambatta G, Baculi F, Hickman M, LeBrun L, Pagarigan B, Carmel G, Lu CC, Lu G, Riley M, Satoh Y, Schafer P, Daniel TO, Carmichael J, Cathers BE, Chamberlain PP. A Cereblon Modulator (CC-220) with Improved Degradation of Ikaros and Aiolos. J Med Chem. 2018 Jan 25;61(2):535-542. doi: 10.1021/acs.jmedchem.6b01921. Epub 2017 Apr 20. PMID 28425720
- [Background] Burtis CA, Ashwood ER. Tietz Textbook of Clinical Chemistry, 3rd ed. Philadelphia; WB Saunders, 1998.